CLINICAL TRIAL: NCT06699433
Title: Utilizing Artificial Intelligence-driven Virtual Standardized Pediatric Patients to Enhance the Capabilities of Primary Healthcare Doctors in China for Managing Common Pediatric Diseases: a Randomized Controlled Trial
Brief Title: Artificial Intelligence-driven Virtual Standardized Pediatric Patients Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Dr. Huanyuan Luo, Professor, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Virtual pediatric patients
Record Dates: First submitted 2024-11-01; First posted 2024-11-21 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pneumococcal Pneumonia; Rotavirus Enteritis With Hypovolemic Shock; Hand-foot-and-mouth Disease; Acute Appendicitis; Respiratory Failure (Pediatric Patients)
MeSH Terms: conditions — Pneumonia, Pneumococcal; Hand, Foot and Mouth Disease; Appendicitis; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual standardized patients (VSPs) training (Experimental): Virtual standardized patients (VSPs), utilizing internet and virtual simulation technology, emulate patients with specific disease characteristics and clinical manifestations. With advantages in safety, flexibility, convenience, and efficiency, VSPs are used in medical education, clinical reasoning training, and licensure examinations. Doctors will interact with VSPs to conduct clinical simulations and training, including consultations, physical examinations, auxiliary examinations, and treatment decision-making, to enhance their capabilities for managing common pediatric diseases
  Interventions: Behavioral: Virtual standardized patients (VSPs)
- Case teaching manuals (Experimental): Doctors will use case teaching manuals to enhance their capabilities for managing common pediatric diseases
  Interventions: Behavioral: Case teaching manuals
- Case teaching videos (Experimental): Doctors will use case teaching videos to enhance their capabilities for managing common pediatric diseases
  Interventions: Behavioral: Case teaching videos

INTERVENTIONS:
Behavioral: Virtual standardized patients (VSPs) — Virtual standardized patients (VSPs), utilizing internet and virtual simulation technology, emulate patients with specific disease characteristics and clinical manifestations. With advantages in safety, flexibility, convenience, and efficiency, VSPs are used in medical education, clinical reasoning training, and licensure examinations. Doctors will interact with VSPs to conduct clinical simulations and training, including consultations, physical examinations, auxiliary examinations, and treatment decision-making, to enhance their capabilities for managing common pediatric diseases
  Arms: Virtual standardized patients (VSPs) training
Behavioral: Case teaching manuals — Doctors will use case teaching manuals to enhance their capabilities for managing common pediatric diseases
  Arms: Case teaching manuals
Behavioral: Case teaching videos — Doctors will use case teaching videos to enhance their capabilities for managing common pediatric diseases
  Arms: Case teaching videos

SUMMARY:
Background: China's healthcare system for children faces significant challenges, particularly due to the limited pediatric service capacity of primary healthcare institutions. A shortage of effective and accessible training tools for primary care doctors further hinders progress in addressing this gap. Technological advancements, especially in artificial intelligence, offer a potential solution to improve pediatric care. Artificial intelligence-driven virtual standardized patients (VSPs), leveraging internet and virtual simulation technologies, simulate clinical cases with specific disease characteristics, providing an innovative, efficient, and flexible training method. VSPs are increasingly utilized in medical education, clinical reasoning, and licensure exams. This study focuses on using VSPs to improve the management of common pediatric conditions, which are major health concerns for children and impose significant psychological and financial burdens on families.

Methods: This study will involve a three-arm randomized controlled trial to evaluate the effectiveness of a virtual pediatric standardized patient platform in enhancing primary care doctors' management of common pediatric diseases. At least 459 participants, including general practitioners, internal medicine practitioners, surgeons, and pediatricians from more than 10 provinces across China, will be randomly assigned to one of three groups: the virtual patient platform group, the case teaching manual group, or the case teaching video group. Five virtual patient cases covering pneumococcal pneumonia, rotavirus enteritis with hypovolemic shock, hand-foot-and-mouth disease, acute appendicitis, and respiratory failure will be developed, along with corresponding case teaching materials. After a two-week learning period, participants' disease management abilities will be assessed using clinical vignettes. The primary outcome is adherence to best clinical practice guidelines, categorized into full adherence, partial adherence, and nonadherence.

Discussion: This study aims to leverage artificial intelligence for capacity enhancement, targeting the shortcomings of primary care pediatrics and using VSP to help enhance primary care pediatrics capacity. It is a randomized controlled trial involving over 300 primary healthcare institutions across more than 10 provinces in China, ensuring broad and representative participation from both developed and underdeveloped regions.

ELIGIBILITY:
1. Inclusion and Exclusion Criteria for Research Institutions

   Inclusion Criteria:
   * Primary and secondary hospitals
   * Community health centers (stations) and clinics, as well as township health centers and village health clinics

   Exclusion Criteria:
   * Specialized medical institutions (such as specialized hospitals and dental clinics)
   * Public health prevention and treatment institutions (such as tuberculosis prevention centers)
   * Ethnic medicine institutions (such as Mongolian and Tibetan hospitals)
   * Hospitals above the secondary level
   * Hospitals that have not yet been graded (due to their short establishment time and potentially unstable operations)
2. Inclusion and exclusion criteria for research subjects

Inclusion Criteria:

* Practicing (assistant) doctors and rural doctors working in medical institutions that meet the above conditions
* With a scope of practice only including general practice, internal medicine, surgery, and pediatrics

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 459 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Doctor adherence to best clinical practice guidelines | Through study completion, an average of 6 months
  Doctor adherence to best clinical practice guidelines, i.e., the extent to which doctors consistently make judgments and treatments based on best clinical practice guidelines and progression of the disease. Ordered categorical variable, consisting of three grades: full adherence, partial adherence, and nonadherence. It will be measured using clinical vignette method.

SECONDARY OUTCOMES:
Dichotomous variable of doctor adherence to best clinical practice guidelines | Through study completion, an average of 6 months
  Dichotomous variable of doctor adherence to best clinical practice guidelines. Dichotomous variable, consisting of two categories: full adherence, partial adherence or no adherence. It will be measured using clinical vignette method.
The degree of accuracy of a doctor's diagnosis according to best clinical practice guidelines | Through study completion, an average of 6 months
  The degree of accuracy of a doctor's diagnosis according to best clinical practice guidelines. Ordered categorical variable, consisting of three categories: fully correct, partially correct, incorrect. It will be measured using clinical vignette method.
Doctor score of examination that is directly related to handling the disease | Through study completion, an average of 6 months
  Doctor score of examination that is directly related to handling the disease. It is a continuous variable. It will be measured using examination paper called Disease Handling Capacity Scale. The lowest score is 0, the highest score is 5, and higher scores mean a better outcome.
Doctor score of examination that is related to expansion skills of handling the disease | Through study completion, an average of 6 months
  Doctor score of examination that is related to expansion skills of handling the disease. It is a continuous variable. It will be measured using examination paper called Expanded Disease Handling Capacity Scale. The lowest score is 0, the highest score is 5, and higher scores mean a better outcome.
The level at which the doctor focuses on meeting the actual needs of the patient and gives due consideration to the patient's feelings | Through study completion, an average of 6 months
  The level at which the doctor focuses on meeting the actual needs of the patient and gives due consideration to the patient's feelings. It is a continuous variable. It will be measured using team-developed patient-centered situational question test paper method.
Adoption of training by doctors | Through study completion, an average of 6 months
  Implementation outcome: Adoption of training by doctors. Dichotomous variable, consisting of two categories: adopted, not adopted. It will be measured using team-developed questionnaire (self-reported by doctors).
Costs to researchers of developing and implementing three types of training | Through study completion, an average of 6 months
  Implementation outcome: Costs to researchers of developing and implementing three types of training. It is a continuous variable. It will be measured using project final account of expenditure.
Doctor score of acceptability of three types of training | Through study completion, an average of 6 months
  Implementation outcome: Doctor score of acceptability of three types of training. It is a continuous variable. It will be measured using generic Theoretical Framework of Acceptability (TFA)-based questionnaire self-reported by doctors.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, Doctor, Principal Investigator — National Clinical Research Center for Child Health and Disorders, Chongqing, China
Locations (3):
- China (3):
  - Yuntan Street Community Health Center, Guiyang, Guizhou
  - Jinxi County People's Hospital, Fuzhou, Jiangxi
  - Honghe County People's Hospital, Yisa, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication, are to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
Access Criteria: All collected IPDs will be provided in a timely manner to anyone who has a valid reason for requesting data from the corresponding author.